CLINICAL TRIAL: NCT01449773
Title: Effects of N-3 Polyunsaturated Fatty Acids On Chylomicron Secretion And Expression Of Genes That Regulate Intestinal Lipid Metabolism In Men With Type 2 Diabetes
Acronym: DBB48
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Patrick Couture, Professor, Laval University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: INAF-117.05.01
Record Dates: First submitted 2011-10-06; First posted 2011-10-10 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- n-3 PUFAs (Experimental)
  Interventions: Dietary Supplement: n-3 PUFAs
- Corn and soybean oil pill (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: n-3 PUFAs — 5 capsules/day in order to provide 3 g/day of n-3 PUFAs.
  Arms: n-3 PUFAs
Dietary Supplement: Placebo — 5 capsules/day containing corn and soybean oil
  Arms: Corn and soybean oil pill

SUMMARY:
The overaccumulation of apoB-48-containing lipoproteins of intestinal origin seen in patients with type 2 diabetes are now thought to be attributable to elevated intestinal production and reduced clearance. Substantial evidence exists indicating that elevated plasma levels of these lipoproteins are associated with increased cardiovascular disease risk. Therefore, reduction of atherogenic plasma triglyceride-rich lipoproteins (TRL) levels of intestinal origin appears to be crucial to improve CVD risk associated with type 2 diabetes. In this regard, n-3 PUFAs have been shown to exert beneficial effects on diabetic dyslipidemia. However, the investigators understanding of the physiological changes that occur with n-3 PUFA supplementation is suboptimal, thereby limiting the investigators appreciation of its impact on CVD risk associated with type 2 diabetes. The effects of n-3 PUFAs on the intestinal production of TRLs and the expression of genes regulating intestinal lipid absorption and chylomicron synthesis have not yet been examined in humans. The general objective of the proposed research is to investigate the mechanisms by which n-3 PUFAs beneficially modify intestinal lipoprotein metabolism in patients with type 2 diabetes. The investigators hypothesize that n-3 PUFA supplementation in men with type 2 diabetes will:

* reduce TRL apoB-48 production rate and increase fractional catabolic rate of these lipoproteins,
* decrease the expression of genes that regulate intestinal lipid absorption and synthesis as well as synthesis of apoB-48-containing lipoproteins,
* decrease both plasma surrogates of cholesterol absorption and cholesterol synthesis.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 55 years,
* plasma TG levels above the 50th percentile for age,
* non-smoker,
* BMI between 25.0 and 40.0 kg/m2,
* stable body weight for at least 6 months prior to the study baseline,
* HbA1c between 6.5 and 8.5%,
* baseline fasting plasma glucose < 15.0 mmol/L
* patients with de novo type 2 diabetes not taking oral hypoglycemic agents -- - or patients having received stable doses of metformin for at least 3 months before randomization.

Exclusion Criteria:

* extreme dyslipidemias such as familial hypercholesterolemia,
* patients with secondary form of diabetes or acute metabolic diabetic complications,
* patients having received or being treated with insulin or a thiazolidinedione within the past 6 months,
* subjects having CVD (CHD, cerebrovascular disease or peripheral arterial disease)
* subjects taking medications known to affect lipoprotein metabolism (e.g. steroids, beta blockers, thiazide diuretics, lipid lowering agents,
* significant alcohol intake

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-04; Primary Completion 2009-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in the in vivo kinetics of intestinally derived apoB-48-containing lipoproteins between the two 8-week interventions | At the end of the two 8-week interventions

SECONDARY OUTCOMES:
Change in the expression of genes that regulate intestinal lipid absorption (NPC1L1, ABCG5/8, FABP, SREBP-1c) and synthesis (DGAT, ACAT2, HMG CoA reductase) as well as synthesis of apoB-48-containing lipoproteins (MTP)between the two 8-week interventions | At the end of the two 8-week interventions
Change in the plasma surrogates of cholesterol absorption (campesterol, beta-sitosterol) and synthesis (lathosterol) between the two 8-week interventions | At the end of the two 8-week interventions

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Couture, MD, PhD, FRCP, Principal Investigator — Laval University
Locations (1):
- Laval University, Québec, Quebec, Canada

REFERENCES:
- [Derived] Labonte ME, Couture P, Tremblay AJ, Hogue JC, Lemelin V, Lamarche B. Eicosapentaenoic and docosahexaenoic acid supplementation and inflammatory gene expression in the duodenum of obese patients with type 2 diabetes. Nutr J. 2013 Jul 15;12:98. doi: 10.1186/1475-2891-12-98. PMID 23855973